CLINICAL TRIAL: NCT00885183
Title: Adjuvant Acupuncture Care for Breast Cancer Patients Experiencing Side Effects From Chemotherapy. A Randomised Controlled Pilot and Feasibility Study
Brief Title: Adjuvant Acupuncture Care for Breast Cancer Patients Experiencing Side Effects From Chemotherapy
Acronym: Acubreast
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficult to recruit participants
Sponsor: University Hospital of North Norway (Other)
Collaborators: Norwegian Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: REK NORD 77/08
Record Dates: First submitted 2009-04-19; First posted 2009-04-21 (Estimated); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Breast Cancer
Keywords: breast cancer; chemotherapy; adjuvant therapy; acupuncture; fatigue; Early stage breast cancer patients
MeSH Terms: conditions — Breast Neoplasms; Fatigue | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- acupuncture therapy (Experimental): Breast cancer patients are randomised to additional 12 acupuncture treatment sessions while undergoing standard chemotherapy
  Interventions: Procedure: Acupuncture therapy
- Usual care (Other): Control group (usual care) receives standard chemotherapy alone
  Interventions: Procedure: Acupuncture therapy

INTERVENTIONS:
Procedure: Acupuncture therapy — 12 acupuncture treatment sessions for a period of 16 weeks

SUMMARY:
Breast cancer patients report many symptoms while undergoing conventional care, including nausea/vomiting, fatigue, pain, depression and anxiety. Existing interventions to address these common side effects of treatment are limited. Patients diagnosed with cancer frequently seek complementary medicine (CAM), and there is a need to investigate potential effects of CAM therapies. This phased pilot and feasibility study has two aims:

1. Develop an acupuncture treatment protocol for adjuvant acupuncture care for breast cancer patients undergoing chemotherapy using structured interviews with established acupuncture teams in Norway.
2. Implement the treatment protocol in a pilot study to evaluate outcome measures, effect sizes and acceptability of acupuncture care delivered alongside conventional care.

Study results will support the design of future research; including a Phase III randomised controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Females, 18 years or older with early stage breast cancer, no previous chemotherapy and no metastatic disease

Exclusion Criteria:

* Needle phobia, use of anticoagulant drugs, inability to comply with study regimen

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-04; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Fatigue scale | Weeks 16 and 29

SECONDARY OUTCOMES:
Health related quality of life: EORTC QLQ-C30, EORTC QLQ-BR23, MYCaw | Weeks 16, 19 and 29
Hospital anxiety and depression scale (HADS) | Weeks 16, 19 and 29

CONTACTS AND LOCATIONS:
Overall Officials: Sameline Grimsgaard, MD, MPH, PhD, Principal Investigator — Clinical Research Centre, University Hospital of North Norway
Locations (1):
- University Hospital of North Norway, Tromsø, Norway